CLINICAL TRIAL: NCT01382654
Title: Two Formulations and Concentrations of Epinastine Nasal Spray Versus Azelastine Nasal Solution for Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 033-102; 033-102 (Other: Inspire Pharmaceuticals)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — epinastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- epinastine 0.1% (Experimental): nasal spray 2 sprays to each nostril for a total of 3 doses
  Interventions: Drug: epinastine 0.1%
- epinastine 0.1% with taste masking agent (Experimental): nasal spray 2 sprays to each nostril for a total of 3 doses
  Interventions: Drug: epinastine 0.1% with taste masking agent
- epinastine 0.2% (Experimental): nasal spray 2 sprays to each nostril for a total of 3 doses
  Interventions: Drug: epinastine 0.2%
- epinastine 0.2% with taste masking agent (Experimental): nasal spray 2 sprays to each nostril for a total of 3 doses
  Interventions: Drug: epinastine 0.2% with taste masking agent
- azelastine 0.1% (Active Comparator): nasal spray 2 sprays in each nostril for a total of 3 doses
  Interventions: Drug: azelastine 0.1%

INTERVENTIONS:
Drug: epinastine 0.1% — nasal spray 2 sprays to each nostril for a total of 3 doses
  Arms: epinastine 0.1%
Drug: epinastine 0.1% with taste masking agent — nasal spray 2 sprays to each nostril for a total for a 3 doses
  Arms: epinastine 0.1% with taste masking agent
Drug: epinastine 0.2% — nasal spray 2 sprays to each nostril for a total of 3 doses
  Arms: epinastine 0.2%
Drug: epinastine 0.2% with taste masking agent — nasal spray 2 sprays to each nostril for a total of 3 doses
  Arms: epinastine 0.2% with taste masking agent
Drug: azelastine 0.1% — nasal spray 2 sprays to each nostril for a total of 3 doses
  Arms: azelastine 0.1%

SUMMARY:
The objectives of this study were to:

* Examine the tolerability of two formulations and two dose concentrations of epinastine.
* Select formulation(s) of epinastine for future studies by evaluating the individual sensory attribute scores of the Nasal Spray Evaluation Questionnaire (NSEQ) collected after each study drug administration and the subject preference ranking assessed at the completion of the study.
* Compare the preference of two formulations and two dose concentrations of epinastine compared to azelastine following a single dose of each in a randomized, double-blind, two-cohort, three-period crossover design.

ELIGIBILITY:
Inclusion Criteria:

* between ages 18-70
* history of SAR or PAR for 1 year
* mild symptoms

Exclusion Criteria:

* asthma or RAD
* respiratory tract infection within 14 days prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Overall preference rank at the completion of the study using the Overall Nasal Spray Evaluation Questionnaire (NSEQ) | 2 days

SECONDARY OUTCOMES:
Scores from each individual response from the NSEQ of all administered formulations (two formulations and two concentrations of epinastine and azelastine). | 2 days